CLINICAL TRIAL: NCT03316573
Title: A Phase 2 Study of Pembrolizumab in Patients With Histiocyte/Dendritic Cell Neoplasms and Biologically Selected Subtypes of Relapsed/Refractory Aggressive Lymphomas
Brief Title: Pembrolizumab in Neoplasms or Lymphomas
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Eric Jacobsen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-448
Record Dates: First submitted 2017-10-18; First posted 2017-10-20 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Histiocytic Sarcoma; Follicular Dendritic Cell Sarcoma; Interdigitating Dendritic Cell Sarcoma
Keywords: Lymphoma; Histiocyte sarcoma; Follicular Dendritic Cell Sarcoma; Interdigitating dendritic cell sarcoma
MeSH Terms: conditions — Lymphoma; Histiocytic Sarcoma; Dendritic Cell Sarcoma, Follicular; Dendritic Cell Sarcoma, Interdigitating | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab will be administered intravenously every 3 weeks for 35 cycles
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — The study drug is an antibody that targets a molecule called PD-1. Blocking PD-1 allow the immune system to attack the cancer more effectively.
  Other Names: Keytruda

SUMMARY:
This research study is studying a drug called pembrolizumab as a possible treatment for aggressive lymphoma or a histiocyte or dendritic cell neoplasm.

The drug involved in this study is:

-Pembrolizumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved pembrolizumab for this specific disease but it has been approved for other uses.

The study drug is an antibody that targets a molecule called programmed cell death protein 1 (PD-1). PD-1 is used to turn down the immune system. In general, this is used by the body to prevent the immune system from being too active. However, several cancers appear to use this pathway to prevent the immune system from attacking them. The theory behind this study is that by blocking PD-1, we may be able to prevent the cancer from hiding from the immune system and allow the immune system to attack the cancer more effectively. There is evidence that the type of lymphoma the participant have may use PD-1 to escape the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Histologically confirmed diagnosis of a histiocyte/dendritic cell neoplasm or relapsed/refractory aggressive lymphoma with at least one of the following features (with review required at a participating study center):

  * Diffuse large B cell lymphoma with Epstein-Barr virus (EBV) positive tumor cells (defined as positive EBV-encoded RNA in tumor cells)
  * Plasmablastic lymphoma
  * T cell/histiocyte rich DLBCL
  * EBV+ T cell lymphoma of any histology; note, patients with angioimmunoblastic T cell lymphoma will be eligible regardless of EBV status
  * Histiocytic sarcoma
  * Follicular dendritic cell sarcoma
  * Interdigitating dendritic cell sarcoma
* For patients with histiocytic sarcoma, interdigitating dendritic cell sarcoma, or follicular dendritic cell sarcoma only: disease that is not amenable to surgical resection and/or radiation therapy with curative intent.
* For lymphoma patients only: At least one prior systemic chemotherapy including an alkylating agent and anthracycline (unless contraindicated), and an anti-cluster of differentiate 20 (CD20) monoclonal antibody if the tumor is CD20+.
* For lymphoma patients only: Participants must have received and relapsed after autologous stem cell transplantation (ASCT), or be ineligible for ASCT (including on the basis of refractory disease), or have declined ASCT
* Age 18 years or older at the time of signing consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Karnofsky ≥70%, see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1,000/microliter (mcL)
  * platelets ≥75,000/mcL (> 30,000 if there is bone marrow involvement with lymphoma)
  * total bilirubin < 1.5 times the institutional upper limit of normal (ULN) OR direct bilirubin < the normal in subjects with total bilirubin >1.5 times the ULN
  * Aspartate aminotransferase (AST)(SGOT)/ alanine aminotransferase (ALT) (SGPT) ≤2.5 × institutional ULN or < 5 times ULN in patients with known hepatic involvement with lymphoma
  * albumin > 2.5 mg/dl
  * creatinine < 1.5 times the normal upper institutional limit OR creatinine clearance ≥60 mL/min/1.73 m2 in participants with creatinine levels > 1.5 times the normal upper institutional limit
  * International normalized ratio (INR), activated partial thromboplastin time (aPTT) or prothrombin time (PT) < 1.5 times the ULN unless subject is receiving anticoagulation therapy as long as PT or aPTT are within therapeutic range of intended use of anticoagulant
* Be willing to provide tissue from a newly obtained core needle or excisional biopsy. Newly-obtained is defined as a specimen obtained up to and including 90 days prior to treatment day 1. Subjects for whom newly obtained samples cannot be provided may be enrolled only with agreement by the overall PI.
* No prior allogeneic transplant unless all of the following apply:

  * At least 5 years from time of transplant
  * Absence of clinically significant graft-versus-host disease (GVHD)
  * Not on immune suppression
  * Approval of overall PI
* Not a candidate for potentially curative therapy at the time of enrollment
* Measurable disease per the Lugano criteria.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 5.4.3 - Contraception for the course of the study through 120 days after the last dose of study medication.
* Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section 5.4.3- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* The effects of pembrolizumab on the developing human fetus are unknown. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Prior treatment with a PD-1, PD-L1 or PD-L2 inhibitor
* Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study day 1 or has not recovered (i.e., < grade 1 or at baseline) from adverse events due to a previously administered agent.
* Participants who have had chemotherapy, targeted small molecule therapy, or radiotherapy within 2 weeks prior to study day 1 (6 weeks for nitrosoureas or mitomycin C) or who has not recovered (i.e., < grade 1 or at baseline) from adverse events due to previously administered agents. Note: subjects with < grade 2 peripheral neuropathy are an exception to this criterion and may qualify for the study.
* Radiation therapy within 2 weeks of study treatment
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a known history of active tuberculosis
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has an active infection requiring systemic therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with the use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal her pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a diagnosis of immunodeficiency or is receiving any form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment or is taking chronic systemic steroids (in doses exceeding 10 mg daily of prednisone equivalent) within 7 days prior to the first dose of trial treatment. Note: Subjects with asthma or chronic obstructive pulmonary disease that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections are not excluded from the study.
* Has a history of non-infectious pneumonitis that required systemic corticosteroid treatment or has active pneumonitis.
* Known active central nervous system involvement and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Active hepatitis B (e.g., hepatitis B surface antigen reactive) or hepatitis C (e.g., hepatitis C virus RNA detectable).
* Human immunodeficiency virus (HIV 1/2).
* Is pregnant or breast-feeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit until 120 days after the last dose of trial treatment.
* Has received a live vaccine within 30 days of planned start of study therapy. (Note: seasonal influenza vaccines for injection are allowed as they are inactivated; however, intranasal influenza vaccines are live attenuated vaccines and are NOT allowed)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab.
* Baseline pulse oximetry <94% or requires oxygen supplementation of any kind
* If subject underwent major surgery they must have recovered adequately from the toxicity and/or complications from the procedure prior to starting therapy.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2026-03-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griffin GK, Weirather JL, Roemer MGM, Lipschitz M, Kelley A, Chen PH, Gusenleitner D, Jeter E, Pak C, Gjini E, Chapuy B, Rosenthal MH, Xu J, Chen BJ, Sohani AR, Lovitch SB, Abramson JS, Ishizuka JJ, Kim AI, Jacobson CA, LaCasce AS, Fletcher CD, Neuberg D, Freeman GJ, Hodi FS, Wright K, Ligon AH, Jacobsen ED, Armand P, Shipp MA, Rodig SJ. Spatial signatures identify immune escape via PD-1 as a defining feature of T-cell/histiocyte-rich large B-cell lymphoma. Blood. 2021 Mar 11;137(10):1353-1364. doi: 10.1182/blood.2020006464. PMID 32871584

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 66 [33 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants]
  00 - Fully active, able to carry on all pre-disease performance without restriction | 6
  01 - Restricted in physically strenuous activity but ambulatory and able to carry out light work | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The number of subjects with partial response (PR) or complete response (CR) by PET/CT scan
  Per Lugano criteria, CR is defined as positron emission tomography-computed tomography (PET-CT), score 1, 2, or 3 with or without a residual mass on 5 point scale (5PS) OR on CT, target nodes/nodal masses must regress to ≤1.5 cm in longest diameter (LDi). PR is defined as PET-CT score 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size. OR on CT ≥50% decrease in the sum of the products of the longest perpendicular diameters (SPD) of up to 6 target measurable nodes and extranodal sites.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 18
Participants | 3

2. Secondary Outcome: Complete Response Rate
Description: The number of patients with complete response (CR)
  Per Lugano criteria, CR is defined as PET-CT, score 1, 2, or 3 with or without a residual mass on 5PS OR on CT, target nodes/nodal masses must regress to ≤1.5 cm in LDi.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 18
Participants | 3

3. Secondary Outcome: Number of Patients With Adverse Events of Any Grade
Description: The number of patients with an adverse event of any grade that has definite, probable, or possible attribution to study treatment.
Time Frame: Up to 35 cycles of treatment (approximately 2 years) plus up to an additional 24 months of follow-up after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 18
Participants | 18

4. Secondary Outcome: Duration of Response
Description: Length of first complete (CR) or partial response (PR) until progression (PD)
  Per Lugano criteria, CR is defined as PET-CT, score 1, 2, or 3 with/without a residual mass on 5PS OR on CT, target nodes/nodal masses must regress to ≤1.5 cm in LDi. PR is defined as PET-CT score 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size. OR on CT ≥50% decrease in SPD of up to 6 target measurable nodes and extranodal sites. PD is defined as PET-CT score 4 or 5 with an increase in intensity of uptake from baseline and/or new fluoro-2-deoxy-D-glucose (FDG)-avid foci consistent with lymphoma at interim or end-of-treatment assessment. OR on CT, an individual node/lesion must be abnormal. OR new/clear progression of pre-existing nonmeasured lesions. OR regrowth of previously resolved lesions. OR new node >1.5 cm in any axis or new extranodal site >1.0 cm in any axis or be unequivocal and attributable to lymphoma. AND/OR new/recurrent involvement of the bone marrow
Time Frame: Up to 35 cycles of treatment (approximately 2 years) plus up to an additional 24 months of follow-up after treatment
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 3
months | 15 [4 to 26]

5. Secondary Outcome: Progression-free Survival
Description: Time from study registration until the earlier of first progression or death from any cause, censored for patients alive without progression or lost to follow-up without documented progression.
  Per Lugano criteria, progression is defined as PET-CT score 4 or 5 with an increase in intensity of uptake from baseline and/or new FDG-avid foci consistent with lymphoma at interim or end-of-treatment assessment. OR on CT, an individual node/lesion must be abnormal. OR new or clear progression of pre-existing nonmeasured lesions. OR regrowth of previously resolved lesions. OR a new node >1.5 cm in any axis or a new extranodal site >1.0 cm in any axis or be unequivocal and must be attributable to lymphoma. AND/OR new or recurrent involvement of the bone marrow
Time Frame: Up to 35 cycles of treatment (approximately 2 years) plus up to an additional 24 months of follow-up after treatment
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 18
months | 1.5 [0.5 to 28]

6. Secondary Outcome: Duration of Complete Response
Description: The length of first complete response (CR) until progression (PD)
  Per Lugano criteria, CR is defined as PET-CT, score 1, 2, or 3 with or without a residual mass on 5PS OR on CT, target nodes/nodal masses must regress to ≤1.5 cm in LDi. PD is defined as PET-CT score 4 or 5 with an increase in intensity of uptake from baseline and/or new FDG-avid foci consistent with lymphoma at interim or end-of-treatment assessment. OR on CT, an individual node/lesion must be abnormal. OR new or clear progression of pre-existing nonmeasured lesions. OR regrowth of previously resolved lesions. OR a new node >1.5 cm in any axis or a new extranodal site >1.0 cm in any axis or be unequivocal and must be attributable to lymphoma. AND/OR new or recurrent involvement of the bone marrow
Time Frame: Up to 35 cycles of treatment (approximately 2 years) plus up to an additional 24 months of follow-up after treatment
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 3
months | 12 [0 to 24]

7. Secondary Outcome: Overall Survival
Description: Time from study registration until death from any cause, censored for patients still alive or lost to follow-up
Time Frame: Up to 35 cycles of treatment (approximately 2 years) plus up to an additional 24 months of follow-up after treatment
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 18
months | 24 [1 to 35]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all patients who received any amount of study treatment from initiation of treatment for up to 35 cycles (approximately 2 years) plus up to an additional 24 months of follow-up after treatment
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 10/18
Serious Adverse Events (participants affected / at risk) | 8/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=18)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Death NOS (General disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — diplopia (double vision)
Hypertension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=18)
Anemia (Blood and lymphatic system disorders) | 10 (29)
Fatigue (General disorders) | 10 (12)
Alkaline phosphatase increased (Investigations) | 9 (15)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (17)
Platelet count decreased (Investigations) | 7 (13)
Nausea (Gastrointestinal disorders) | 7 (8)
White blood cell decreased (Investigations) | 6 (18)
Aspartate aminotransferase increased (Investigations) | 6 (16)
Alanine aminotransferase increased (Investigations) | 6 (10)
Diarrhea (Gastrointestinal disorders) | 6 (8)
Neutrophil count decreased (Investigations) | 5 (21)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 4 (15)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Fever (General disorders) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Chills (General disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Lymphocyte count decreased (Investigations) | 3 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (8)
Sinus tachycardia (Cardiac disorders) | 3 (5)
Headache (Nervous system disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (3) — Mouth pain, Ventral hernia, Oral bleeding
Hyperthyroidism (Endocrine disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2) — Pancytopenia, Lymphocytopenia
Hypertension (Vascular disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (4)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (4) — Transaminitis, Hepatotoxicity, Transaminitis, Transaminitis
Hypokalemia (Metabolism and nutrition disorders) | 1 (3)
Weight loss (Investigations) | 1 (2)
Wound infection (Infections and infestations) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Iritis
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Rigors
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Pneumonia
Infusion related reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Erythematous Rash
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03316573/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03316573/ICF_001.pdf